CLINICAL TRIAL: NCT02733289
Title: Standard Follow-up Program Cervix Cancer (SFP CERVIX)
Acronym: SFPCERVIX
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: 201600207
Record Dates: First submitted 2016-03-17; First posted 2016-04-11 (Estimated); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Cervical Cancer Radiation Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years

SUMMARY:
Standard evaluation and follow-up data regarding complications of curative radiation treatment for cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* Every cervical cancer patient with curative intent for radiotherapy, treated at our department

Exclusion Criteria:

* Non-curative treatment
* Part of the treatment is given in another hospital

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Every patient who receives curative radiotherapy for cervical cancer at the department of Radiotherapy at the UMCG.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2015-06; Primary Completion 2040-12 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
Complications | Five years
  Physiological parameters, questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Jannet Beukema, Principal Investigator — Principal Investigator
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands